CLINICAL TRIAL: NCT04933760
Title: CV-SQuISH-ED: A Clinical Validation Solving the Question of Inflammation or Sepsis Hastily in the Emergency Department
Brief Title: CV-SQuISH-ED: Clinical Validation Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cytovale, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CV-CLN-007
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Sepsis; Infection
Keywords: Sepsis
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Cytovale IntellipSep test — The Cytovale IntelliSep test measures a series of physical properties that indicate activation of leukocytes obtained from a venous K2-EDTA anti-coagulated whole blood sample.

SUMMARY:
This is a study to evaluate the diagnostic performance of the investigational Cytovale System & IntelliSep Test as a diagnostic marker of sepsis in a population of patients presenting to the emergency department with signs or suspicion of infection compared to retrospective physician adjudication, per the sepsis 3 definition, of those patients.

DETAILED DESCRIPTION:
This is a multi-site prospective study to evaluate the diagnostic performance of the investigational Cytovale System & IntelliSep Test for patients presenting to the Emergency Department with signs or suspicion of infection. The IntelliSep Test is a microfluidic test that measures the biophysical properties of human leukocytes in conjunction with other laboratory findings and clinical assessments to aid in the early detection of sepsis with organ dysfunction occurring within the first three days after the blood sample collection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. The first vital sign (any one of: blood pressure, temperature, pulse or respiratory rate) has been recorded in the medical record
3. A 300µl blood sample originally collected in a K2 EDTA (hematology purple top) tube within 4 hours of the first recorded vital sign is available.
4. Sign or suspicion of infection, defined as meeting either of criterion A-1 and A-2 (based on temperature, WBC, heart rate, respiratory rate and/or culture order criteria):

Exclusion Criteria:

1. Patients in whom a palliative care or hospice course is expected during ED visit
2. Self-reported, documented or otherwise known to be actively enrolled on any experimental/investigational therapeutic medication prior to blood collection
3. Self-reported, documented, or known history of a hematologic malignancy (any leukemia, lymphoma, or myeloma), myelodysplastic syndrome, or myeloproliferative disorder
4. Self-reported, documented or otherwise known to receive a chemotherapeutic agent or other excluded medication in the past 3 months (Appendix C)
5. Self-reported, documented or otherwise known to have undergone a hematopoietic stem cell transplant or any solid organ transplant
6. Patients transferred to the Emergency Department from another acute care facility
7. Residents or patients of a hospital-based skilled nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Emergency Department with signs or suspicion of infection.
Sampling Method: Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
IntelliSep Index versus Retrospective Physician Diagnosis (RPD) per the sepsis 3 definition | 30 days
  To validate the diagnostic performance of the investigational Cytovale System & IntelliSep Test as a diagnostic marker of sepsis in a population of patients presenting to the emergency department with signs or suspicion of infection, the IntelliSep test score is compared to the non-reference method of retrospective physician adjudication, per the sepsis 3 definition, of those patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya Jagneaux, MD, Principal Investigator — Lady of the Lake Regional Medical Center; Hariharan Regunath, MD, Principal Investigator — University of Missouri-Columbia; Liza Rosenman, MD, Principal Investigator — University of Washington; Simon Mahler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - University of Missouri, Columbia, Missouri
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No